CLINICAL TRIAL: NCT06656351
Title: B-FREE Chronic Babesiosis Study: A Phase 2 Open Label Study of Tafenoquine for Treatment of Chronic Babesiosis Patients With Severe Fatigue
Brief Title: B-FREE Chronic Babesiosis Study
Acronym: TQ-BA-2024-3
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: 60 Degrees Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQ-BA-2024-3
Record Dates: First submitted 2024-10-22; First posted 2024-10-24 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Chronic Babesiosis
Keywords: Chronic Babesiosis
MeSH Terms: interventions — tafenoquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tafenoquine (Experimental): Tafenoquine (2 x 100 mg tablets) will be self-administered orally with food on Days 1, 2, 3, 4, then weekly thereafter for a total 12-week treatment period. Weekly treatment will start on Day 11 and end on Day 89.
  Interventions: Drug: Tafenoquine 100mg

INTERVENTIONS:
Drug: Tafenoquine 100mg — Tafenoquine

SUMMARY:
Phase 2 Open Label Study of Tafenoquine for Treatment of Chronic Babesiosis Patients with Severe Fatigue

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged ≥ 18 years
* Severe disabling fatigue
* Have at least one common symptom of babesiosis
* Have laboratory evidence of exposure to babesia in the last 12 months
* Able and willing to give written informed consent
* Able and willing to perform all study assessments
* If female negative urine pregnancy test and
* If female agree to use an acceptable method of birth control

Exclusion Criteria:

* Glucose-6-phosphate-dehydrogenase (G6PD) deficiency
* Breastfeeding
* Unmanaged Psychotic disorder
* Known hypersensitivity reaction to tafenoquine or other 8-aminoquinolines
* Current or planned treatment with quinine
* Uncontrolled cardiopulmonary or endocrine disorders
* Taking OCT2/MATE substrates without appropriate medical oversight
* Medical history of chronic, active viral diseases including HIV/AIDS, hepatitis B, and hepatitis C
* Have a risk factors for relapsing babesiosis
* Anorexia
* Any concomitant significant illness unrelated to babesiosis
* The patient is unable to tolerate medication by the oral route
* The patient has previously taken tafenoquine
* Hemoglobin at baseline is ≤ 8 g/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change in General Fatigue | From enrollment until Day 90 of treatment.
  The Multidimensional Fatigue Inventory (MFI) is a 20-item, patient-reported scale. designed to evaluate five dimensions of fatigue: general fatigue (items 1, 5, 12, 16), physical fatigue (items (items 2, 8, 14, 20), reduced motivation (items 3, 6, 10, 17), reduced activity (items 4, 9, 15, 18), and mental fatigue (items 7, 11, 13, 19) (Smets-1995). Items are scored 1-5, with 10 positively phrased items reverse scored (items 2, 5, 9, 10, 13, 14, 16, 17, 18, 19). This scale has been used to assess treatment outcomes in patients with chronic fatigue syndrome, women with fibromyalgia, Parkinson's disease, patients undergoing anti-cancer treatment, and the impact of fatigue on the quality of life in rheumatoid arthritis. Total scale score, and each of the 5 subscales scores will be calculated. MFI subscales are scored by summing four items, each has five possible responses giving a range of possible scores from 4 to 20.

SECONDARY OUTCOMES:
Babesia nucleic acid test (NAT) | From baseline until Day 90 of treatment.
  Percentage of patients achieving molecular cure at or earlier than Day 90 who tested positive on the Babesia NAT at baseline, with molecular cure defined as the observance of a negative Babesia NAT test on or before Day 90
Babesia nucleic acid test (NAT) | From baseline until Day 90 of treatment
  Proportion of patients with a reactive NAT test at baseline who had a non-reactive NAT test at Day 90
Babesia nucleic acid test (NAT) and RT PCR | From baseline, Days 30, 60, 90, 120, and 180
  Number and percentage of patients with a negative Babesia screen on Days 30, 60, 90, 120, and 180 who tested positive at baseline, as assessed individually for each molecular diagnostic test (rtPCR, dPCR, and NAT)

CONTACTS AND LOCATIONS:
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No